CLINICAL TRIAL: NCT05639829
Title: Time-restricted Eating in Survivors Trial
Acronym: TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HREBA.CC-20-0077
Record Dates: First submitted 2022-11-09; First posted 2022-12-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-11

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weekday time-restricted eating (Experimental): The intervention consisted of 8 weeks of ad libitum TRE with a 12-8 pm 8-hour eating window on weekdays. Participants received instructions to only consume water, black coffee, or black tea from 8 pm to 12 pm on weekdays and during the weekend, where there were no restrictions on eating timing. No other dietary or physical activity instructions were given.
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — Restriction of calorie intake to an 8-hour window, with water only fasting in the remaining 16 hours of the 24-hour period
  Other Names: intermittent fasting

SUMMARY:
Breast cancer survivors aged 60+ and with overweight/obesity who had completed chemotherapy 1-6 years earlier completed 8 weeks of 12-8 pm weekday-only time-restricted eating. The intervention was delivered by a registered dietitian call, twice-daily automated text messages asking about eating start/stop times, and three support phone calls.

ELIGIBILITY:
Inclusion Criteria:

* history of early-stage (I-III) breast cancer
* completed anthracycline-based chemotherapy 1-6 years earlier
* aged ≥60 years
* had a body mass index (BMI) >25 kg/m2

Exclusion Criteria:

* taking lipid, glucose, or weight-lowering medications
* contraindications to maximal exercise testing or research MRI
* unstable thyroid disorder
* self-reported history of an eating disorder
* self-reported diagnosis of type 1 or 2 diabetes
* weight loss of ≥15 lbs in previous 3 months
* working night shifts
* could not provide consent in English

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Framingham 10-year cardiovascular risk score (%) | 8 weeks
  Calculated using the Canadian Cardiovascular scoring system

SECONDARY OUTCOMES:
Visceral adipose tissue | 8 weeks
  measured via magnetic resonance fat-water separation imaging
Thigh adipose tissue fraction | 8 weeks
  Relative measure of amount of inter+intra muscular adipose tissue within the thigh muscle measured via magnetic resonance fat-water separation imaging
Liver adipose tissue fraction | 8 weeks
  Relative measure of amount of adipose tissue within the liver
Cardiorespiratory fitness | 8 weeks
  Measured as peak volume of oxygen consumed collected with a cycle erogmeter exercise test
Resting energy expenditure | 8 weeks
  Collected via metabolic cart in supine resting position after overnight fast
Respiratory quotient | 8 weeks
  Collected via metabolic cart in supine resting position after overnight fast
Lipid profile | 8 weeks
  Collected via analysis of fasting blood sample by Lifelabs commercial laboratory
Hemoglobin A1c | 8 weeks
  Collected via analysis of blood sample by Lifelabs commercial laboratory
Waist circumference | 8 weeks
  measured as the average of two measurements to the nearest 0.5 cm.
Fasting glucose | 8 weeks
  Collected via analysis of fasting blood sample by Lifelabs commercial laboratory
Fasting insulin | 8 weeks
  Collected via analysis of fasting blood sample by Lifelabs commercial laboratory
Resting systolic and diastolic blood pressure | 8 weeks
  measured as the average of two measurements 60 seconds apart following 5-10 minutes of supine rest using an automated device
Body mass | 8 weeks
  measured by physicians scale after overnight fast
Whole-body fat mass | 8 weeks
  estimated using8-point bioelectric impedance (Seca)
Whole-body fat-free mass | 8 weeks
  estimated using8-point bioelectric impedance (Seca)

OTHER OUTCOMES:
Dietary intake | 8 weeks
  Measured via diet records on 3 consecutive weekdays that were analyzed via Food Processor Nutrition Analysis Software
Activity | Change between measurement at baseline and 8 weeks
  24-hour Measured via Sensewear Pro accelerometer worn on the arm for 3 consecutive weekdays
Adherence to intervention | Ongoing for duration of intervention
  Collected via participant responses to automated text messages asking participants to self-report the time they started and stopped eating each day. Calculated as the % of prescribed days to follow the intervention where participant reported performing a 16 hour or longer fast.
Participant acceptability | 8 weeks
  assessed by a researcher-developed end of study questionnaire as: 1) a subjective difficulty rating for following TRE on a scale of 1-10 and 2) rating the dietitian and support calls as 'very helpful' or 'somewhat helpful' on a 5-point Likert scale (other options were 'neutral,' 'somewhat helpful,' and 'unhelpful')
Intervention fidelity | 8 weeks
  determined as completion rates of the intervention components (registered dietitian consult call, the three support calls, and response rate to the text messages)
Intervention sustainability | 1 month post intervention
  Rate of continuing to follow TRE one-month post-intervention completion (without further support or instructions) collected by phone follow-up
Intervention sustainability confidence | 8 weeks
  Average subjective rating of confidence, on 0-100% scale, in ability to follow TRE for one year or longer
Intervention delivery cost | Through study completion, lasting 12-24 weeks depending on chemotherapy protocol
  Estimated as average time spent by personnel on intervention delivery multiplied by the hourly rate for that personnel
Symptoms | Through study completion, lasting 12-24 weeks depending on chemotherapy protocol
  Collected at each of the support phone calls at weeks 1, 3, 6 of the intervention. The research coordinator asked participants if they experienced any symptoms on a pre-determined list or any additional symptoms. Symptoms were only recorded if the participant reported that they were related to the intervention or were unsure if they were related. Symptoms attributed to other life events (i.e., heat wave, stress at work) were not recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Edmonton Clinic Health Academy, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No